CLINICAL TRIAL: NCT01212718
Title: Stratified and Randomized Multi-center Phase II - to Determine Potential Benefit of Treating Patients With Advanced Colorectal Cancer According to the Intratumoral TS RNA Levels
Brief Title: Response Prediction in Metastasized Colorectal Cancer Using Intratumoral Thymidylate Synthase
Acronym: FOGT5
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Ulm (Other)
Collaborators: Pfizer, Berlin Germany (Unknown); Medac, Hamburg, Germany (Unknown); Study Group Oncology of Gastrointestinal Tumors (FOGT) (Unknown)
Responsible Party: Prof. Dr. Marko Kornmann, University of Ulm
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FOGT5
Record Dates: First submitted 2010-09-09; First posted 2010-10-01 (Estimated); Last update posted 2010-10-01 (Estimated); Status verified 2010-09

CONDITIONS: Colorectal Cancer; Non Resectable Metastasis; Reference Lesion; Biopsy; Thymidylate Synthase Quantitation
Keywords: Colorectal Cancer; non resectable metastasis; reference lesion; biopsy; thymidylate synthase quantitation
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Neoadjuvant Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 5-FU (Active Comparator): FUFA 5-flurouracil and folinic acid control
  Interventions: Drug: FUFA
- Folfiri (Active Comparator): 5-fluouracil and folinic acid in combination with irinotecan (Folfiri) systemic chemotherapy intensified treatment arm
  Interventions: Drug: systemic chemotherapy

INTERVENTIONS:
Drug: FUFA — 2600/500 mg/m2 i.v. 24 h via port, 1 time weekly for six weeks, than have a break for 2 weeks (=8 weeks for 1 cycle)
  Arms: 5-FU
Drug: systemic chemotherapy — CPT-11, 80 mg/m2 for 90 minutes and 5 FU/FA 2000/500 mg/m2 iv. 24h via port; 1 time weekly for six weeks, than have a break for 2 weeks
  Arms: Folfiri

SUMMARY:
The aim of the study was to evaluate the feasibility of TS determination in a multicenter trial setting using a central facility for measurement and confirm its role as predictive factor for 5-FU treatment in MCRC.

DETAILED DESCRIPTION:
Eligible were patients with non-resectable metastasized or recurrent histologically proven CRC with the presence of a reference lesion two-dimensional measurable and accessible for a biopsy.The biopsy was taken from the reference lesion either by surgery during primary tumor resection, by trans-cutaneous true-cut needle biopsy or by trans-anal approach. Intratumoral relative TS mRNA expression levels were determined using samples shipped in RNA-preserving solution or as glass slides after microdissection of tumor cells. An independent company stratified the patients according to ther relative TS mRNA expression level in TS low and TS high followed by randomization to receive either FUFA of Folfiri. Response to chemotherapy was evaluated and documented according to the RECIST criteria after every therapy cycle.

ELIGIBILITY:
Inclusion Criteria:

* patients (>= 18 years) with non-resectable metastasized or recurrent histologically proven CRC with the presence of a reference lesion two-dimensional measurable and accessible for a biopsy
* a performance status WHO 0-2 (Karnofsky >= 60%)
* an estimated life expectancy of at least 3 months
* written informed consent

Exclusion Criteria:

* patients older than 75 years not fulfilling these criteria
* brain metastases or a secondary cane
* a history of a systemic palliative chemotherapy
* and an adjuvant chemotherapy (within 6 months)
* pregnant or nursing women
* a known allergy toward irinotecanhydroclorid or of any ingredients of Campto or other severe medical
* laboratory and social conditions not allowing chemotherapy and follow-up

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Actual)
Dates: Start 2001-07; Primary Completion 2010-06 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Best response to first-line chemotherapy (recist) | 1 year
  Response to chemotherapy was evaluated and documented according to the RECIST criteria after every therapy cycle (every two months).

SECONDARY OUTCOMES:
overall survival, toxicity, treatment related complications, time to progression | 3-year
  See above.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of General, Visceral, and Transplantations Surgery, Univeristy of Ulm, Ulm, Germany